CLINICAL TRIAL: NCT02015494
Title: Phase 1 Study of the Safety and Immunogenicity of VAX2012Q: A Quadrivalent Influenza Vaccine in Healthy Adults Age 18-40 Years
Brief Title: Phase 1 Safety Study of Recombinant Influenza Vaccine for Prevention
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: VaxInnate Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VAX2012Q-01; BARDA (Other Grant/Funding Number: HHSO10020110011C)
Record Dates: First submitted 2013-12-09; First posted 2013-12-19 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Influenza
Keywords: Safety; Immunogenicity
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- 4 mcg VAX2012Q (Experimental): 4 mcg VAX2012Q
  Interventions: Biological: VAX2012Q
- 8 mcg VAX2012Q (Experimental): 8 mcg VAX2012Q
  Interventions: Biological: VAX2012Q
- 14 mcg VAX2012Q (Experimental): 14 mcg VAX2012Q
  Interventions: Biological: VAX2012Q
- 18 mcg VAX2012Q (Experimental): 18 mcg VAX2012Q
  Interventions: Biological: VAX2012Q
- 12 mcg VAX2012Q (Experimental): 12 mcg VAX2012Q
  Interventions: Biological: VAX2012Q
- 8 mcg VAX2012Q repeated (Experimental): 8 mcg VAX2012Q
  Interventions: Biological: VAX2012Q
- 12 mcg VAX2012Q repeated (Experimental): 12 mcg VAX2012Q
  Interventions: Biological: VAX2012Q

INTERVENTIONS:
Biological: VAX2012Q — Recombinant influenza HA vaccine delivered IM
  Other Names: Quadrivalent Recombinant Hemagglutinin Influenza vaccine

SUMMARY:
One dose of escalating strengths of an investigational influenza vaccine VAX2012Q (Quadrivalent Recombinant Hemagglutinin Seasonal Influenza Vaccine) will be evaluated for tolerability and immunogenicity in healthy adults 18-40 years of age.

DETAILED DESCRIPTION:
This is a multi-center, open-label, dose escalating study in which up to 320 healthy subjects age 18-40 years will be administered VAX2012Q at one of up to 7 dose levels. VAX2012Q vaccine will be formulated at the clinical site ("field mix") from the four components (VAX128C, VAX181, VAX173 and VAX172) in diluent to produce ten doses in a multi-dose vial for use within 12 hours of preparation. The dose will be prepared from appropriate dilutions from the monovalent drug product vials. Data for safety and immunogenicity will be collected after each dose with safety being assessed after each dose level and immune response, after dose level 4. Reactogenicity and safety labs through Day 1 will be reviewed by the Safety Monitoring Committee (SMC) prior to enrolling in the next dose level.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18-40 years of age at the time of vaccination in good health as determined by medical history, physical exam, laboratory assessments and the clinical judgment of the Principal Investigator
* Able to provide informed consent indicating that they understand the purpose of this study and are willing to adhere to the procedures described in this protocol
* If the subject is a female of childbearing potential, she must use adequate contraceptive precautions (e.g., intrauterine contraceptive device, oral contraceptives or other equivalent hormonal contraception) for 2 months prior to vaccination and continue to use such precautions for a minimum of three months after vaccination. She must also have a negative urine pregnancy test within 24 hours prior to receiving study vaccine. Women at least one year post-menopausal or surgically sterile will not be considered of childbearing potential.
* Willing to receive the unlicensed vaccine given as an IM injection
* Willing to provide multiple blood specimens collected by venipuncture

Exclusion Criteria:

* Use of any investigational or non-registered drug or vaccine product within 30 days preceding the administration of the study vaccine or planned use within the first six weeks of the study period
* Has received any licensed or other investigational influenza vaccine within 3 months prior to enrollment in this study or expected receipt of any influenza vaccination before the Day 21 blood collection
* History of excessive alcohol use, drug abuse or significant psychiatric illness
* Tobacco use within 3 months of enrollment and throughout first 6 months of the study
* Has a chronic illness (e.g., liver or kidney disease), receiving a concomitant therapy or have any other condition that could interfere with the subject's participation in the study or in the interpretation of the study results
* Clinically significant abnormal liver function tests at screening
* Positive serology for HBsAg, HCV or HIV antibodies
* Pregnant or lactating female
* Having cancer or have received treatment for cancer within three years (persons with a history of cancer who are disease-free without treatment for three years or more are eligible), excluding minor skin cancers, which are allowed unless located at the vaccination site
* Persons with impaired immune responsiveness (of any cause), including diabetes mellitus and autoimmune disorders
* Persons presently receiving or having a recent history of receiving (within the past six months) any medication or therapeutic modality that affects the immune system such as allergy shots, immune globulin, interferon, immunomodulators, radiation therapy, cytotoxic drugs or drugs known to be frequently associated with significant major organ toxicity, or systemic corticosteroids (oral or injectable). Inhaled and topical corticosteroids are allowed.
* Persons with a history of severe allergic reaction after previous vaccinations or hypersensitivity to any seasonal influenza vaccine component
* Persons with a history of Guillain-Barré Syndrome
* Receipt of blood or blood products 8 weeks prior to vaccination or planned administration during the three week study period following vaccination
* Donation of blood or blood products within 8 weeks prior to vaccination or during the three week study period following
* An oral temperature >100.4° or acute disease within 72 hours prior to vaccination, defined as the presence of a moderate or severe illness (as determined by the investigator through medical history and physical examination; for example, those requiring an absence from work) with or without fever.
* Body Mass Index >29.9
* Any disorder of coagulation
* A clinical diagnosis of influenza within the previous 12 months
* Any other condition or circumstance which, in the opinion of the Principal Investigator, poses an unacceptable risk for participation in the study

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 316 (Actual)
Dates: Start 2014-03; Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Safety | 21 Days
  Injection site and systemic symptoms will be collected for 21 days after vaccination. Other AEs assessed as related to vaccination will be collected at a 6 month clinic visit and a 1 year phone call.

SECONDARY OUTCOMES:
Immunogenicity | 21 days and 6 months post-vaccination
  Immune response to vaccine will be measured by serum HAI levels

CONTACTS AND LOCATIONS:
Overall Officials: C. Jo White, MD, Study Director — VaxInnate Corporation
Locations (4):
- United States (4):
  - Johnson County Clin-Trials, Lenexa, Kansas
  - Rochester Clinical Research, Inc, Rochester, New York
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Tekton Research, Austin, Texas

REFERENCES:
- [Background] Taylor DN, Treanor JJ, Strout C, Johnson C, Fitzgerald T, Kavita U, Ozer K, Tussey L, Shaw A. Induction of a potent immune response in the elderly using the TLR-5 agonist, flagellin, with a recombinant hemagglutinin influenza-flagellin fusion vaccine (VAX125, STF2.HA1 SI). Vaccine. 2011 Jul 12;29(31):4897-902. doi: 10.1016/j.vaccine.2011.05.001. Epub 2011 May 17. PMID 21596084
- [Background] Treanor JJ, Taylor DN, Tussey L, Hay C, Nolan C, Fitzgerald T, Liu G, Kavita U, Song L, Dark I, Shaw A. Safety and immunogenicity of a recombinant hemagglutinin influenza-flagellin fusion vaccine (VAX125) in healthy young adults. Vaccine. 2010 Dec 6;28(52):8268-74. doi: 10.1016/j.vaccine.2010.10.009. Epub 2010 Oct 20. PMID 20969925